CLINICAL TRIAL: NCT01506700
Title: Real Time Optical Coherence Tomography (OCT) of Human Tissue
Status: Terminated | Type: Observational
Why Stopped: additional recruitment not needed
Sponsor: Diagnostic Photonics, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: DXP 2012-01
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optical Coherence Tomography — Optical coherence tomography will be used to image tissue structure on excised and in vivo specimens.

SUMMARY:
This is a single-arm, prospective, study of an optical imaging device on approximately twenty (20) subjects undergoing lumpectomies at one study site. In vivo and ex vivo imaging will be performed on study subjects with results being compared to final pathology.

DETAILED DESCRIPTION:
This study is a single-center, prospective, two-part open label study of an optical imaging device on approximately twenty (20) subjects at one (1) study site. Patients scheduled to undergo a lumpectomy will be recruited by the clinical investigators at the investigational site in accordance with the inclusion and exclusion criteria. The study period per subject is the time it takes to assess the in vivo and ex vivo breast tissue samples using the study device during their lumpectomy.

All specimens will be marked with India ink and undergo standard post-operative histology, and digital histology images corresponding to the inked locations will be obtained. The images and the matched digitized post-operative histology images will then be randomized and read by a blinded, independent pathologist. Sensitivity and specificity will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older
2. Signed ICF
3. Women who have been histologically diagnosed with invasive ductal carcinoma or invasive lobular carcinoma of the breast prior to surgery
4. Planning breast preservation
5. Patients undergoing lumpectomy (partial mastectomy) procedure

Exclusion Criteria:

1. Multicentric disease (histologically diagnosed cancer in two different quadrants of the breast)
2. Neoadjuvant systemic therapy
3. All T4 tumors
4. Previous radiation in the operated breast
5. Prior surgical procedure in the same quadrant
6. Implants in the operated breast
7. Pregnancy
8. Lactation
9. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of Optical Coherence Tomography to identify whether or not tumor can be identified ex vivo on breast cancer specimens as compared to post-surgical histology conclusions. | One week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Boppart, MD, PhD, Study Chair — University of Illinois and Diagnostic Photonics, Inc.
Locations (1):
- Carle Foundation Hospital, Urbana, Illinois, United States